CLINICAL TRIAL: NCT00566696
Title: A Reduced Intensity Conditioning Regimen With CD3-Depleted Hematopoietic Stem Cells to Improve Survival for Patients With Hematologic Malignancies Undergoing Haploidentical Stem Cell Transplantation
Brief Title: Mismatched Family Member Donor Transplantation for Children and Young Adults With High Risk Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFLEX; NCI-2011-03670 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2016-05-03 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2019-10

CONDITIONS: Leukemia, Acute Lymphocytic (ALL); Leukemia, Myeloid, Acute(AML); Leukemia, Myeloid, Chronic(CML); Juvenile Myelomonocytic Leukemia (JMML); Hemoglobinuria, Paroxysmal Nocturnal (PNH); Hodgkin Lymphoma; Lymphoma, Non-Hodgkin (NHL); Myelodysplastic Syndrome (MDS)
Keywords: Haploidentical stem cell transplant; Allogeneic stem cell transplant; Mismatched family member stem cell donor transplant; Bone marrow transplant; High risk hematologic malignancies; T cell depletion methodology; Miltenyi Biotec CliniMACS stem cell selection device; Campath-1H intravenous
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Juvenile; Hemoglobinuria; Hemoglobinuria, Paroxysmal; Hodgkin Disease; Lymphoma; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes | interventions — Stem Cell Transplantation; fludarabine; fludarabine phosphate; Thiotepa; Melphalan; Mycophenolic Acid; Rituximab; Alemtuzumab; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Granulocyte Colony-Stimulating Factor; Filgrastim; Muromonab-CD3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-Risk Hematologic Malignancies (Experimental): Participants meeting eligibility criteria undergo haploidentical stem cell transplantation along with systemic chemotherapy and antibodies, including Fludarabine, Thioplex®, L-phenylalanine mustard, mycophenolate mofetil, CellCept®, Rituxan™, Muromonab (prior to January 2010) or Alemtuzumab (after January 2010), Cyclophosphamide, Anti-thymocyte globulin (Rabbit), and G-CSF.
  Grafts from suitable haploidentical donors are processed using the CliniMACS system.
  Interventions: Device: CliniMACS; Procedure: Stem cell transplantation; Drug: Fludarabine; Drug: Thioplex®; Drug: L-phenylalanine mustard; Drug: Mycophenolate mofetil; Drug: Rituxan™; Drug: Alemtuzumab; Drug: Cyclophosphamide; Drug: Anti-thymocyte globulin (Rabbit); Drug: G-CSF; Drug: Muromonab

INTERVENTIONS:
Device: CliniMACS — Miltenyi Biotec CliniMACS stem cell selection device
Procedure: Stem cell transplantation — An infusion of HLA mismatched family member donor stem cells processed through the use of the investigational Miltenyi Biotec CliniMACS device.
Drug: Fludarabine — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Fludara
Drug: Thioplex® — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Thiotepa; TESPA; TSPA
Drug: L-phenylalanine mustard — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Melphalan; Phenylalanine mustard; L-PAM; L-sarcolysin; Alkeran
Drug: Mycophenolate mofetil — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: MMF; CellCept®
Drug: Rituxan™ — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Rituximab
Drug: Alemtuzumab — After January 2010, due to the unavailability of muromonab, transplant recipients received a conditioning regimen consisting of systemic chemotherapy and antibodies, including alemtuzumab.
  Other Names: Campath-1H; Campath®
Drug: Cyclophosphamide — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Cytoxan
Drug: Anti-thymocyte globulin (Rabbit) — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Thymoglobulin®; Rabbit ATG
Drug: G-CSF — Transplant recipients will receive a conditioning regimen consisting of systemic chemotherapy and antibodies.
  Other Names: Filgrastim; Neupogen®
Drug: Muromonab — Prior to January 2010, transplant participants received a conditioning regimen consisting of systemic chemotherapy and antibodies, including muromonab. Muromonab became unavailable from the manufacturer at that time and was replaced by alemtuzumab.
  Other Names: OKT3; Muromonab-CD3

SUMMARY:
Blood and marrow stem cell transplant has improved the outcome for patients with high-risk hematologic malignancies. However, most patients do not have an appropriate HLA (immune type) matched sibling donor available and/or are unable to identify an acceptable unrelated HLA matched donor through the registries in a timely manner. Another option is haploidentical transplant using a partially matched family member donor.

Although haploidentical transplant has proven curative in many patients, this procedure has been hindered by significant complications, primarily regimen-related toxicity including GVHD and infection due to delayed immune reconstitution. These can, in part, be due to certain white blood cells in the graft called T cells. GVHD happens when the donor T cells recognize the body tissues of the patient (the host) are different and attack these cells. Although too many T cells increase the possibility of GVHD, too few may cause the recipient's immune system to reconstitute slowly or the graft to fail to grow, leaving the patient at high-risk for significant infection.

For these reasons, a primary focus for researchers is to engineer the graft to provide a T cell dose that will reduce the risk for GVHD, yet provide a sufficient number of cells to facilitate immune reconstitution and graft integrity. Building on prior institutional trials, this study will provide patients with a haploidentical (HAPLO) graft engineered to specific T cell target values using the CliniMACS system. A reduced intensity, preparative regimen will be used in an effort to reduce regimen-related toxicity and mortality.

The primary aim of the study is to help improve overall survival with haploidentical stem cell transplant in this high risk patient population by 1) limiting the complication of graft versus host disease (GVHD), 2) enhancing post-transplant immune reconstitution, and 3) reducing non-relapse mortality.

DETAILED DESCRIPTION:
This study will explore the following objectives:

1. To assess if the event-free survival at one-year post-transplant for research participants with high-risk hematologic malignancies can be improved following HAPLO hematopoietic stem cell transplant (HSCT) using a graft depleted of CD3+ cells ex vivo and a reduced intensity-conditioning regimen.

Secondary objectives:

1. To estimate the one-year overall survival (OS) and disease-free survival (DFS) for research participants who receive this study treatment.
2. To estimate the cumulative incidence of relapse for research participants who receive this study treatment.
3. To estimate the rate of overall grade III-IV acute GVHD, and the rate and severity of chronic GVHD in research participants.
4. To estimate the incidence of non-hematologic regimen-related toxicity and regimen-related mortality in the first 100 days post-transplant.

Exploratory objectives:

1. To explore the biologic significance of soluble interleukin-2 receptor and immunologic state [quantitative lymphocyte studies, V beta spectratyping, T-cell receptor excision circles (TREC) assay] to predict the development of acute and chronic GVHD in these research participants.
2. To measure the pharmacokinetics of Campath-1H in pediatric HAPLO HSCT recipients

NOTE: This protocol originally used muromonab (OKT3) in the conditioning regimen to prepare participants for haploidentical HCT. After muromonab became unavailable from the manufacturer in 2010, muromonab was replaced by alemtuzumab (Campath-1H) for use in subsequent participants.

ELIGIBILITY:
Inclusion Criteria:(transplant recipient)

* Patients less than or equal to 21 years of age; may be greater than 21 years old if a current St. Jude patient or previously treated St. Jude patient within 3 years of completion of prior treatment.
* Must have one of the following diagnosis:

  * ALL high risk in second remission. Examples include relapse on therapy, first remission duration of less than or equal to 30 months, or relapse within 12 months of completing therapy.
  * ALL in third or subsequent remission.
  * ALL high risk in first remission. Examples include: induction failure, minimal residual disease greater than or equal to 1% marrow blasts by morphology after induction, persistent or recurrent cytogenetic or molecular evidence of disease during therapy requiring additional therapy after induction to achieve remission.
  * High-risk AML in first remission. Examples include monosomy 7, M6, M7, t(6;9), FLT3-ITD, or patients who have greater than or equal to 25% blasts by morphology after induction or who do not achieve CR after 2 courses of therapy (includes myeloid sarcoma).
  * Relapsed or persistent AML (less than or equal to 25% blasts in marrow by morphology).
  * AML in second or subsequent morphologic remission (includes myeloid sarcoma).
  * CML in first chronic phase with detectable molecular or cytogenetic evidence of disease despite medical therapy; or CML with a history of accelerated or blast crisis, now in chronic phase; or unable to tolerate tyrosine kinase inhibitor therapy.
  * Juvenile myelomonocytic leukemia (JMML).
  * Myelodysplastic syndrome (MDS).
  * Therapy related (secondary) AML, ALL, or MDS.
  * Hodgkin lymphoma after failure of prior autologous HSCT or unsuitable for autologous HSCT.
  * Non-Hodgkin lymphoma (NHL) in second complete remission (CR2) or subsequent.
* Has not received a prior allogeneic hematopoietic stem cell transplant.
* Does not have a suitable HLA-matched sibling donor available for stem cell donation.
* Does not have a suitable cord blood product or volunteer matched unrelated donor (MUD) available in the necessary time for stem cell donation.
* Has a suitable HLA partially matched family member available for stem cell donation.
* Cardiac shortening fraction greater than or equal to 25%.
* Creatinine clearance or glomerular filtration rate (GFR) greater than or equal to 40 ml/min/1.73 m^2.
* Forced vital capacity (FVC) greater than or equal to 40% of predicted value or a pulse oximetry value of greater than or equal to 92% on room air.
* Direct bilirubin less than or equal to 3 mg/dl.
* Age-dependent performance score of greater than or equal to 50.
* Serum glutamic pyruvic transaminase (SGPT) less than 3 times the upper limit of normal for age.
* Karnofsky or Lansky (age-dependent) performance score of greater than or equal to 50.
* No known allergy to murine products or human anti-mouse antibody (HAMA) results within normal limits.
* Not pregnant (confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment).
* Not breast feeding.

Inclusion criteria (stem cell donor):

* Partially HLA matched family member.
* At least 18 years of age.
* Human immunodeficiency virus (HIV) negative.
* Not pregnant (confirmed by negative serum or urine pregnancy test within 7 days prior to enrollment).
* Not breast feeding.

Inclusion criteria (transplant recipient - stem cell boost)

Has experienced one of the following disorders post-transplant:

* graft failure
* graft rejection
* delayed hematopoietic and/or immune reconstitution.

Exclusion: NA

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2007-12-14 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 73 enrollments at St. Jude Children's Research Hospital between 12/2007 and 12/2013. Of the 73, 37 were non-patient donors who did not receive therapeutic intervention, and therefore, no outcome data was collected.
Groups:
- High-Risk Hematologic Malignancies: Participants meeting eligibility criteria and who underwent haploidentical stem cell transplantation with systemic chemotherapy and antibodies, including Fludarabine, Thioplex®, L-phenylalanine mustard, mycophenolate mofetil, CellCept®, Rituxan™, Muromonab (prior to January 2010) or Alemtuzumab (beginning January 2010), Cyclophosphamide, Anti-thymocyte globulin (Rabbit), and G-CSF.
Period: Overall Study
Arm/Group | High-Risk Hematologic Malignancies
Started | 73
Completed | 31
Not Completed | 42
Not completed — Met Exclusion Criteria | 2
Not completed — Muromonab not available | 1
Not completed — Health Status Change | 1
Not completed — Physician Decision | 1
Not completed — Non-Patient Donors | 37

BASELINE CHARACTERISTICS:
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was evaluated at the time of transplantation.
  years | 13.3 (4.69)
Age, Customized [Median (Full Range); unit: years] — Age was evaluated at the time of transplantation.
  years | 14.2 [3.54 to 20.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 20
  More than one race | 1
  Unknown or Not Reported | 2
Conditioning Drug Received [Number; unit: participants]
  Muromonab (OKT3) | 11
  Alemtuzumab (Campath-1H) | 20

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: To determine if one year event-free survival can be improved in pediatric patients undergoing a haploidentical transplant by using a reduced intensity conditioning regimen and a targeted dose T cell depleted donor product. EFS is defined as time from transplantation to the occurrence of relapse or death due to any cause. Patients who are alive at the time of analysis will be censored. The estimated percentage of participants with EFS at one-year post-transplantation is reported using Kaplan-Meier analysis.
Time Frame: one year post-transplant
Measure: Number; unit: Percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Percentage of participants | 54.8

2. Secondary Outcome: Overall Survival (OS)
Description: Estimate the one-year overall survival (OS) for research participants who receive this study treatment. OS is defined as time from transplantation to death due to any cause. Patient who are alive at the time of analysis will be censored. The estimated percentage of participants with OS at one-year post-transplantation is reported using Kaplan-Meier analysis.
Time Frame: one year post-transplant
Measure: Number; unit: Percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Percentage of participants | 71.0

3. Secondary Outcome: Disease-Free Survival (DFS)
Description: Estimate the one-year disease-free survival (DFS) for research participants who receive this study treatment. DFS is defined as time from transplantation to the occurrence of relapse or death due to relapse. Patients who are alive at the time of analysis or die due to other causes will be censored at the time of their events. The estimated percentage of participants with DFS at one-year post-transplantation is reported using Kaplan-Meier analysis.
Time Frame: One year post-transplant
Measure: Number; unit: Percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Percentage of participants | 70.1

4. Secondary Outcome: Incidence of Non-hematologic Regimen-related Toxicities
Description: Estimate of the incidence of non-hematologic regimen-related toxicity and regimen-related toxicity in the first 100 days post-transplant. The percentage of participants are reported by maximum grade seen using binomial distribution. Participants were graded for toxicity using Common Terminology Criteria for Adverse Events version 3.0. In general, Grade 1 is mild, 2 is moderate toxicity but generally does not require treatment, 3 is severe enough to require treatment, 4 is life-threatening, and 5 means it was associated with death.
Time Frame: 100 days post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
percentage of participants
  Grade 1 | 0
  Grade 2 | 3.2
  Grade 3 | 61.3
  Grade 4 | 19.4
  Grade 5 | 16.1

5. Secondary Outcome: Incidence of Regimen-related Mortality
Description: The incidence of regimen-related mortality in the first 100 days post-transplant is estimated based on binomial distribution.
Time Frame: 100 days post-transplant
Measure: Number; unit: Percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Percentage of participants | 9.68

6. Secondary Outcome: To Estimate the Cumulative Incidence of Relapse for Research Participants Who Receive This Study Treatment.
Description: The Cumulative Incidence of Relapse will be reported as the proportion of number of relapses since transplant to the total number of patients at risk at five years post-transplant.
Time Frame: five years post-transplant
Measure: Number; unit: Percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Percentage of participants
  The Cumulative Incidence of Relapse at five year p | 30.0
  Estimate±SE | 8.6

7. Secondary Outcome: To Estimate the Rate of Overall Grade III-IV Acute GVHD, and the Rate and Severity of Chronic GVHD in Research Participants.
Description: The rate of Overall Grade III-IV Acute AVHD will be report as the proportion of patients who have Grade III-IV Acute GVHD to the total patients with transplant. The rate of Chronic GVHD will be report as the proportion of patients who have Chronic GVHD to the total patients with transplant. The Severity of Chronic GVHD will be reported using CTCAE grading system, as a number.
Time Frame: five years post-transplant
Measure: Number; unit: Percentage of participants
Arm/Group | High-Risk Hematologic Malignancies
Number analyzed (Participants) | 31
Percentage of participants
  Rate of Overall Grade III-IV Acute AVHD | 22.58
  Rate of limited grade Chronic GVHD | 9.68

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of participant enrollment through December 23, 2015.
Arm/Group | High-Risk Hematologic Malignancies
All-Cause Mortality (participants affected / at risk) | 16/31
Serious Adverse Events (participants affected / at risk) | 20/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Risk Hematologic Malignancies (N=31)
Allergic reaction, micafungin (Immune system disorders) | 1 (1)
Graft failure (Blood and lymphatic system disorders) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Post-transplant lymphoproliferative disease (Blood and lymphatic system disorders) | 1 (1)
Fever without neutropenia (General disorders) | 9 (11)
Headache (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Vomiting (disorder) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, diffuse alveolar (Vascular disorders) | 1 (1)
Failure, hepatic (Hepatobiliary disorders) | 1 (1)
Veno-occlusive disease, hepatic (Hepatobiliary disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2)
Adult respiratory distress syndrome (disorder) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Failure, renal (Renal and urinary disorders) | 2 (2)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 4 (5)
Fever without neutropenia (Infections and infestations) | 6 (6)
Hepatitis (Infections and infestations) | 1 (1)
Infection, acinetobacter baumannii, blood (Infections and infestations) | 1 (1)
Infection, aceinetobacter calcoaceticus, baumannii, blood (Infections and infestations) | 1 (2)
Infection, coagulase negative staphylocuccus, skin (Infections and infestations) | 1 (1)
Infection, enterobacter cloacae, blood culture (Infections and infestations) | 1 (1)
Infection, enterococcus faecalis, blood (Infections and infestations) | 1 (1)
Infection, influenza type A, respiratory tract (Infections and infestations) | 1 (1)
Infection, staphylocuccus epidermidis, blood (Infections and infestations) | 1 (4)
Infection, urinary tract, gamma hemolytic streptococcus (Infections and infestations) | 1 (1)
Infection, vancomycin-resistant enterococcus, blood (Infections and infestations) | 1 (1)
Infection, vancomycin resistant enterococcus, blood/Hickman line (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | High-Risk Hematologic Malignancies (N=31)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 6 (8)
Hypotension (Cardiac disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 4 (4)
Nausea (finding) (Gastrointestinal disorders) | 3 (3)
Vomiting (disorder) (Gastrointestinal disorders) | 2 (2)
Epistaxis (Vascular disorders) | 4 (4)
Hemorrhagic cystitis (Vascular disorders) | 2 (2)
Elevated ALT (SGPT) (Metabolism and nutrition disorders) | 3 (3)
Elevated GGT (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (disorder) (Metabolism and nutrition disorders) | 5 (7)
Hypophosphatemia (disorder) (Metabolism and nutrition disorders) | 2 (2)
Confusion (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Hemorrhagic cystitis (Renal and urinary disorders) | 3 (3)
Cytokine Release Syndrome (Campath) [10/20 (50%)] (General disorders) | 10/20 (10) — 20 received Campath and were at risk
Cytokine Release Syndrome (muromonab) [3/11 (27.27%)] (General disorders) | 3/11 (3) — 11 received muromonab and were at risk
Cytokine Release Syndrome (Stem Cell Infusion) (General disorders) | 3 (3)
Headache (General disorders) | 2 (2)
Pain, generalized, multiple sites (General disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 24 (25)
Fever without neutropenia (Infections and infestations) | 2 (2)
Infection, adenovirus, blood (Infections and infestations) | 3 (3)
Infection, adenovirus, respiratory tract (Infections and infestations) | 2 (2)
Infection, adenovirus, stool (Infections and infestations) | 4 (7)
Infection, BK Virus, bladder (Infections and infestations) | 2 (2)
Infection, BK Virus, blood (Infections and infestations) | 8 (9)
Infection, BK Virus, urine (Infections and infestations) | 7 (8)
Infection, Clostridium Difficile, stool (Infections and infestations) | 4 (5)
Infection, herpes simplex, lip (Infections and infestations) | 2 (2)
Infection, Klebsiella pneumoniae, blood (Infections and infestations) | 2 (2)
Infection, vancomycin-resistant enterococcus, rectum (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT00566696/Prot_SAP_000.pdf